CLINICAL TRIAL: NCT05379049
Title: Evaluation of the Therapeutic Response to TNF-alpha Antagonist (Etanercept, Infliximab, Adalimumab) in Patients With Rheumatoid Arthritis; Using Plasma TNF-alpha as a Competent Biomarker. Single Center Study in Sulaymaniyah/ Iraq
Brief Title: Therapeutic Response to Tumor Necrosis Factor-alpha (TNF-alpha) Antagonists in Rheumatoid Arthritis.
Acronym: TNF-alpha
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sulaimani (Other)
Responsible Party: Principal Investigator, Hiwa Khidhir Saaed, Lecturer and researcher at Department of Pharmacology & Toxicology, College of Pharmacy, University of Sulaimani
Other Study IDs: UoS
Record Dates: First submitted 2022-05-07; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis; Inflammatory Arthritis; Ankylosing Spondylitis
Keywords: Rheumatoid Arthritis, Cytokines
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis; Spondylitis, Ankylosing | interventions — Etanercept; Infliximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human Blood:
  CBC (complete blood count), C-reactive protein and ESR as inflammatory biomarkers, and detecting TNF-alpha and IL-6
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Biological: Infliximab: Adalimumab; Etanercept; — Therapeutic drug monitoring, evaluation of clinical outcomes and laboratory analysis of biomarkers
  Other Names: Remicade, Remsima، Humira, amgevita، Enbrel

SUMMARY:
Rheumatoid arthritis (RA) is an autoimmune, chronic inflammatory disease and TNF-alpha has been recognized as a triggering cytokine in the induction of joints inflammation and is involved in the pathogenesis of RA.

Treatment for RA aims to reduce disease activity, prevent or manage joint deterioration and lower the risk of major comorbidities such as heart disease and stroke.

The strategy of targeting cytokines has significantly increased RA patient outcomes. Therefore management with biological disease-modifying antirheumatic drugs "bDMARD" (Etanercept, Infliximab, Adalimumab) should be considered, If the treatment goal is not met with the first conventional synthetic drug modifying antirheumatic drugs (csDMARD) strategy, or if there are poor prognostic factors.

The multi-biomarker disease activity test could be used to help standardise individual treatment decisions, especially in patients who failed to respond well to the traditional treatment.

Iraq does not currently have specific guidelines, which might pose a risk to patients' safety. More data about the choice of bDMARD is needed in terms of tracking therapeutic response, or whether TNF or other pro-inflammatory cytokines like interleukin-6 (IL-6) is the main factor for the development and severity of RA.

These data are important to improve the overall status of the patient, better choice of treatment and biomarkers to detect.

There is limited information on the treatment patterns of rheumatoid arthritis (RA) across Iraq including the Kurdistan Region. Therefore, the aim of this research is to evaluate the efficacy, and clinical responses of RA patients who have been treated with different anti-TNF, as well as on answering the research hypothesis, Can plasma TNF-alpha and IL-6 be used as markers of therapeutic response to TNF alpha antagonist in patients with RA?

DETAILED DESCRIPTION:
Rheumatologists in Iraq, including those in the Kurdistan Region, rely on the European League Against Rheumatism (EULAR) and the American College of Rheumatology (ACR) guidelines and publications due to a lack of evidence-based national guidelines.

Several studies found that targeting TNF-alpha in the early stages of RA and evaluating serum TNF- levels, in combination with DAS28's assessment of disease clinical activity to track disease progression could result be advantageous for patients on anti-TNF medication in the future.

Objectives: The current research focuses on identifying the efficacy of three TNF-alpha antagonists (Etanercept, Infliximab, and Adalimumab) used currently in Sulaymaniyah Hospitals.

Methodology, an observational open-label study of ~60-80 adult patients with active RA from both genders that are registered at Rehabilitation and Rheumatology Center in Sulaymaniyah City who have been treated with biological agents (Etanercept, Infliximab, Adalimumab), regardless of disease activity and concomitant treatments.

Baseline data will be collected during the first visit and patients will be followed up during the study at regular intervals.

The study includes data of patients after filling the patient consent form, and are willingly giving their demographic data such as; Age, Sex, and Race (ethnic group). and answer the questions of multidimensional health assessment. Also measuring patients' weight at each visit, The clinical assessment of the patients is based on DAS28 (Disease Activity Score) by using ESR(Erythrocyte Sedimentation Rate), and VAS (Visual analogue score).

The laboratory data or the biomarkers at each visit include; CBC (complete blood count), C-reactive protein and ESR as inflammatory biomarkers, and detecting TNF-alpha and IL-6 to indicate the efficacy of the treatment and better choice of the treatment.

As for the statistical analysis plan, the Software SPSS (version 27) will be used.

Demographic and nominal results will be reported in percentages and frequencies.

Numerical results will be reported as the mean and standard deviation in cases of normal distribution, and as the median and interquartile range (IQR) in cases of skewed distribution.

The continuous variables CRP, TNF, IL-6 and the change over time, will be analyzed using linear mixed models for repeated measures. The chi-squared test will be used for dichotomous variables.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the ACR/EULAR 2010 criteria for rheumatoid arthritis (RA).
* Patients (or Legal Guardian, if applicable) who are willing to give informed consent for the study period-time follow up.
* Concomitant DMARDs
* Duration of treatment with TNF-alpha antagonists <1 year, 1-5 years, >5 years

Exclusion Criteria:

* Tubercle Bacillus (TB)
* Hepatitis B, Hepatitis C
* Pregnancy and lactation
* Patients with heart failure.
* Previous or concurrent malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ~60-80 adult patients [≥18 years] with Rheumatoid Arthritis from both genders registered at Rehabilitation and Rheumatology Center in Sulaymaniyah City, who are not responding to conventional DMARDs regardless of disease activity and concomitant treatments.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of Plasma Tumor Necrosis Factor alpha (TNF-α) among different TNF alpha antagonist Therapy in Patients with Rheumatoid Arthritis. | Up to 12 Weeks
  Tumor Necrosis Factor alpha (TNF-α) is a pro-inflammatory cytokine produced by activating macrophages and T-cells that play a key role in the production of other cytokines and the induction of chronic inflammation.
Comparison of Plasma Interleukin-6 (IL-6) among different TNF alpha antagonist Therapy in Patients with Rheumatoid Arthritis. | Up to 12 Weeks
  Interleukin-6 (IL-6) is a major pro-inflammatory cytokine, triggers the vicious circle of escalating RA disease activity via inducing immune activation and inflammation in RA.
Mean change of C-reactive Protein (CRP) among different TNF alpha antagonist Therapy in Patients with Rheumatoid Arthritis. | Up to 12 Weeks
  C-reactive protein (CRP) a potential marker of systemic inflammation and is elevated in patients with rheumatoid arthritis (RA).
Mean change of Erythrocyte Sedimentation Rate (ESR) among different TNF alpha antagonist Therapy in Patients with Rheumatoid Arthritis. | Up to 12 Weeks
  Erythrocyte sedimentation rate (ESR) is a popular hematology test that may detect and track an increase in inflammatory activity in the body, which can be caused by autoimmune illness, infections, or malignancies.
Complete blood count (CBC) | Up to 12 Weeks
  A complete blood count (CBC) is a blood test used to evaluate overall health and detect a wide range of hematological disorders, including anemia.
Assessment of Disease Activity Score (DAS) | Up to 12 weeks
  Disease Activity Score (DAS) is a continuous measure of RA disease activity that combines information from swollen joints, tender joints, acute phase response and general health.
Assessment of Visual Activity Score (VAS) | Up to 12 weeks
  Visual Activity Score (VAS) A psychometric pain rating scale for parameters that range across a continuum of values, such as pain. The VAS pain scale ranges from "no pain" to "worst pain," and patients mark a line to indicate how they are feeling.

SECONDARY OUTCOMES:
A correlation between plasma Tumor Necrosis Factor alpha (TNF-α) and disease activity and severity. | Up to 12 weeks
  To determine how different Tumor Necrosis Factor-alpha (TNF-α) antagonist medications affected plasma (TNF-α) levels and the Disease Activity Score (DAS) in rheumatoid arthritis (RA) patients.
A correlation between plasma Interleukin-6 (IL-6) and disease activity and severity. | Up to 12 weeks
  To determine how different Tumor Necrosis Factor-alpha (TNF-α) antagonist medications affected plasma Interleukin-6 (IL-6) levels and the Disease Activity Score (DAS) in rheumatoid arthritis (RA) patients.

CONTACTS AND LOCATIONS:
Overall Officials: Hiwa Saaed, PhD, Principal Investigator — University of Sulaimani College of Pharmacy; Sana M Mohammed, BSc, Principal Investigator — Directorate of Health, Sulaymaniyah
Locations (1):
- Hiwa Khidhir Saaed, Sulaymaniyah, Kurdistan Region, Iraq

IPD SHARING:
Plan to Share IPD: No
The data will be presented as a Mean of the sample population.

REFERENCES:
- [Background] Inam Illahi M, Amjad S, Alam SM, Ahmed ST, Fatima M, Shahid MA. Serum Tumor Necrosis Factor-Alpha as a Competent Biomarker for Evaluation of Disease Activity in Early Rheumatoid Arthritis. Cureus. 2021 May 29;13(5):e15314. doi: 10.7759/cureus.15314. PMID 34221763
- [Background] Smolen JS, Landewe RBM, Bijlsma JWJ, Burmester GR, Dougados M, Kerschbaumer A, McInnes IB, Sepriano A, van Vollenhoven RF, de Wit M, Aletaha D, Aringer M, Askling J, Balsa A, Boers M, den Broeder AA, Buch MH, Buttgereit F, Caporali R, Cardiel MH, De Cock D, Codreanu C, Cutolo M, Edwards CJ, van Eijk-Hustings Y, Emery P, Finckh A, Gossec L, Gottenberg JE, Hetland ML, Huizinga TWJ, Koloumas M, Li Z, Mariette X, Muller-Ladner U, Mysler EF, da Silva JAP, Poor G, Pope JE, Rubbert-Roth A, Ruyssen-Witrand A, Saag KG, Strangfeld A, Takeuchi T, Voshaar M, Westhovens R, van der Heijde D. EULAR recommendations for the management of rheumatoid arthritis with synthetic and biological disease-modifying antirheumatic drugs: 2019 update. Ann Rheum Dis. 2020 Jun;79(6):685-699. doi: 10.1136/annrheumdis-2019-216655. Epub 2020 Jan 22. PMID 31969328
- [Background] Oderda GM, Lawless GD, Wright GC, Nussbaum SR, Elder R, Kim K, Brixner DI. The potential impact of monitoring disease activity biomarkers on rheumatoid arthritis outcomes and costs. Per Med. 2018 Jul 1;15(4):291-301. doi: 10.2217/pme-2018-0001. Epub 2018 Apr 25. PMID 29693487
- [Background] Abbasi M, Mousavi MJ, Jamalzehi S, Alimohammadi R, Bezvan MH, Mohammadi H, Aslani S. Strategies toward rheumatoid arthritis therapy; the old and the new. J Cell Physiol. 2019 Jul;234(7):10018-10031. doi: 10.1002/jcp.27860. Epub 2018 Dec 7. PMID 30536757
- [Background] Xiao Q, Li X, Li Y, Wu Z, Xu C, Chen Z, He W. Biological drug and drug delivery-mediated immunotherapy. Acta Pharm Sin B. 2021 Apr;11(4):941-960. doi: 10.1016/j.apsb.2020.12.018. Epub 2020 Dec 31. PMID 33996408